CLINICAL TRIAL: NCT06862375
Title: Weight Loss Through Mayo Clinic Diet; a Prospective Pilot Study
Brief Title: Weight Loss Through Mayo Clinic Diet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tamim I. Rajjo, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-011982
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mayo Clinic Diet (Experimental): Subjects in the Mayo Clinic Diet (MCD) arm will be provided with options including the Mayo Clinic Diet book 3rd edition or application from digital wellness or both with full subscription paid for by the Mayo Clinic Diet for the 12 week period. The Mayo Clinic Diet arm will switch to usual care after 12 weeks.
  Interventions: Behavioral: Mayo Clinic Diet; Behavioral: Usual Care
- Usual Care (Active Comparator): Subjects in the usual care arm will be provided with two Mayo Clinic resources for lifestyle modifications: Eat Well Use the Plate hand out, and the Food, Physical Activity and Weight Tracking Apps with a list of self-monitoring tools to support a healthy lifestyle. The usual care arm will switch to the Mayo Clinic Diet after 12 weeks.
  Interventions: Behavioral: Mayo Clinic Diet; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Mayo Clinic Diet — Subjects will utilize their choice of the following resources for 12 weeks:
  * Mayo Clinic Diet book, 3rd Edition
  * Digital Wellness app subscription
  * Both the Mayo Clinic Diet book and Digital Wellness app
Behavioral: Usual Care — Subjects will be given the 'Eat Well Use the Plate' informational hand-out, as well as a list of food, physical activity and weight tracking apps to be utilized as resources for self-monitoring .

SUMMARY:
The purpose of study is to evaluate the efficacy of the Mayo Clinic Diet in clinically significant weight loss (>5%) versus usual care. We also wish to evaluate the feasibility, barriers to completion, and sustainability of this intervention at the 24, and 52-week marks. Lastly, we aim to study the change in participants body composition and quality of life at the end of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (non-pregnant) 18-64
* BMI > or = to 25 kg/m2
* Ability to read and understand English. (as the Mayo Clinic Diet book and app are only available in English)

Exclusion Criteria:

* Have a current diagnosis of melanoma or cancer diagnosis
* Currently breastfeeding
* Pregnant, or planned to be pregnant within 6 months
* Have a diagnosis of Type 1 or 2 Diabetes Mellitus
* Had weight loss surgery within the last year
* Currently participating in another lifestyle weight loss program or taking medications for weight loss
* Have lost 5% or more of their weight in the last six months
* Have a history of eating disorders
* Have planned surgery in the next 6 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Mayo Clinic Diet- Was It Worth It survey | 12 weeks, 24 weeks
  The Mayo Clinic Diet - Was It Worth It survey consists of 6 questions to get feedback on the subjects perception of the program.

SECONDARY OUTCOMES:
Mayo Clinic Diet 12-item Short Form health (SF-12) survey | Baseline, 12 weeks, 24 weeks
  The 12-item short form health survey is a self-reported assessment of a subjects health, consisting of physical health and emotional health domains. Emotional health questions are rated on a 5-point Likert scale with 0 = "All of the time" and 5 = "None of the time". Physical health questions are rated on a 3-point Likert scale with 0 = "Yes, Limited A Lot" and 3 = "No, Not Limited At All".

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Rajjo, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials